CLINICAL TRIAL: NCT06826573
Title: Analysis of Risk Factors for High Intraocular Pressure and Retinal Detachment Recurrence After Vitrectomy with Silicone Oil Tamponade in Retinal Detachment Patients
Status: Recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Principal Investigator, Hui Peng, PH.D, First Affiliated Hospital of Chongqing Medical University
Other Study IDs: 2024-130-01
Record Dates: First submitted 2025-02-10; First posted 2025-02-14 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2024-09

CONDITIONS: Rhegmatogenous Retinal Detachment
MeSH Terms: interventions — Intraocular Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- group 1: Subjects who exhibit elevated intraocular pressure during the follow-up period.
  Interventions: Diagnostic Test: Intraocular pressure
- group 2: Subjects with normal intraocular pressure during the follow-up period.
  Interventions: Diagnostic Test: Intraocular pressure
- group 3: Subjects who experience retinal detachment recurrence during the follow-up period.
  Interventions: Diagnostic Test: retinal recovery status
- group 4: Subjects who do not experience retinal detachment recurrence during the follow-up period.
  Interventions: Diagnostic Test: retinal recovery status

INTERVENTIONS:
Diagnostic Test: Intraocular pressure — Intraocular pressure will be measured and recorded at 1 day, 1 week, 1 month, 3 months, 6 months postoperatively, and before silicone oil removal.
  Groups: group 1; group 2
Diagnostic Test: retinal recovery status — Measure and record the retinal recovery status 1 day, 1 week, 1 month, 3 months, 6 months after surgery and before silicone oil removal.
  Groups: group 3; group 4

SUMMARY:
This study is a retrospective study. Patients who visited the ophthalmology clinic of the First Affiliated Hospital of Chongqing Medical University between September 1, 2024, and December 31, 2025, will be screened according to the inclusion and exclusion criteria mentioned below. After obtaining informed consent, clinical data of the subjects will be collected. The surgical procedure will involve "vitrectomy + retinal laser photocoagulation + retinal reattachment + silicone oil tamponade (+ cataract extraction + intraocular lens implantation)." Observation indicators will be recorded at various time points postoperatively: 1 day, 1 week, 1 month, 3 months, 6 months, and before silicone oil removal. Any emergent events occurring during the trial will be treated accordingly. Finally, data will be statistically analyzed to identify risk factors for high intraocular pressure and retinal detachment recurrence in patients with rhegmatogenous retinal detachment.

ELIGIBILITY:
Inclusion Criteria:

* 1. Diagnosed with "rhegmatogenous retinal detachment". 2. Aged over 18 years old, with normal mental and psychological status, regardless of gender.

  3. Intraocular pressure of both eyes is less than 21 mmHg before surgery, and having no personal or family history of glaucoma.

  4. Cup - to - disc ratio (C/D) in fundus examination is less than 0.5 for both eyes.

  5. Those who understand the purpose of this study, sign the "Informed Consent Form" and have a high degree of compliance.

Exclusion Criteria:

- 1. Those with high intraocular pressure before surgery and suffering from ophthalmic diseases such as glaucoma; 3. Those with acute or chronic systemic infections and hematological diseases; 4. Those with a history of mental and psychological diseases; 5. Those with incomplete survey data or unable to cooperate with this research. 5. Those with traumatic rhegmatogenous retinal detachment; 6. Those with active ocular infectious lesions in either eye; 7. Those with severe refractive media opacity (such as corneal nebula, corneal leukoma) in the target eye, which affects imaging examinations during postoperative follow - up.

8. Those with a history of congenital structural abnormalities in the target eye; 9. Those who have undergone vitrectomy for other vitreoretinal diseases in the target eye before screening; 10. Those whom the researchers consider unfit to participate in this clinical trial.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study includes patients with rhegmatogenous retinal detachment who visited the ophthalmology clinic of the First Affiliated Hospital of Chongqing Medical University between September 1, 2024, and December 31, 2025.
Sampling Method: Non-Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Intraocular pressure | The study will be conducted from September 1, 2024, to December 31, 2025. Key follow-up time points include 1 day, 1 week, 1 month, 3 months, 6 months postoperatively, and before silicone oil removal
  If the intraocular pressure is greater than 21 mmHg at any time during the follow - up period, it is considered as an increase in intraocular pressure.
the retinal recovery status | The study will be conducted from September 1, 2024, to December 31, 2025. Key follow-up time points include 1 day, 1 week, 1 month, 3 months, 6 months postoperatively, and before silicone oil removal.
  Measure and record the retinal status 1 day, 1 week, 1 month, 3 months, 6 months after surgery and before silicone - oil removal. If retinal detachment occurs again, it is regarded as the recurrence of retinal detachment.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Our institution has established strict privacy - protection policies. Our organization adheres to high - level data - security regulations. These regulations prohibit the sharing of any patient - related data, including individual patient data, to prevent potential data breaches and ensure the confidentiality of patients' personal and medical information.